| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan (RAP) |
| Title | : | Reporting and Analysis Plan for An Open-Label One-way Interaction Clinical Trial to Evaluate the Pharmacokinetic Interactions Between GSK3640254 and Tenofovir Alafenamide/Emtricitabine in Healthy Subjects |
| <b>Compound Number</b> | ÷ | GSK3640254 |
| <b>Effective Date</b> | : | 29-APR-2019 |

# **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 208134.
- This RAP is intended to describe the full analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | INTRO | DUCTIO | N | 4 |
| 2. | SUMM<br>2.1.<br>2.2.<br>2.3.<br>2.4. | Changes<br>Study Ob<br>Study De | KEY PROTOCOL INFORMATION | 4<br>4<br>5 |
| 3. | PLANN<br>3.1. | | LYSESalyses | |
| 4. | ANALY<br>4.1. | | PULATIONS Deviations | |
| 5. | | ENTIONS<br>Study Tr<br>Baseline<br>Other Co | ONS FOR DATA ANALYSES AND DATA HANDLING S eatment & Sub-group Display Descriptors Definitions onsiderations for Data Analyses and Data Handling ions | 9<br>9 |
| 6. | STUD<br>6.1. | | ATION ANALYSESv of Planned Study Population Analyses | |
| 7. | PHARI<br>7.1. | | Pharmacokinetic Analyses Endpoint / Variables 7.1.1.1. Drug Concentration Measures 7.1.1.2. Derived Pharmacokinetic Parameters Summary Measure Population of Interest Statistical Analyses / Methods 7.1.4.1. Statistical Methodology Specification | 12<br>12<br>12<br>12<br>12 |
| | 7.2. | Seconda<br>7.2.1.<br>7.2.2.<br>7.2.3.<br>7.2.4. | Pharmacokinetic Analyses Endpoint / Variables 7.2.1.1. Drug Concentration Measures 7.2.1.2. Derived Pharmacokinetic Parameters. Summary Measure Population of Interest Statistical Analyses / Methods | 13<br>13<br>13<br>14 |
| 8. | SAFET<br>8.1.<br>8.2.<br>8.3. | Adverse<br>Clinical L | YSES Events Analyses Laboratory Analyses afety Analyses | 15 |
| 9. | REFER | RENCES. | | 16 |
| 10 | APPEN | NDICES | | 17 |

208134

| 10.1. | Appendi | x 1: Schedule of Activities | 17 |
|-------|----------|-----------------------------------------------------|----|
| | 10.1.1. | Protocol Defined Schedule of Events | 17 |
| 10.2. | Appendi | x 2: Study Phases and Treatment Emergent Adverse | |
| | Events | | |
| | 10.2.1. | Study Phases | 21 |
| | | 10.2.1.1. Study Phases for Concomitant Medication | 21 |
| | 10.2.2. | Treatment Emergent Flag for Adverse Events | 22 |
| 10.3. | Appendi | x 3: Data Display Standards & Handling Conventions | |
| | 10.3.1. | Reporting Process | |
| | 10.3.2. | Reporting Standards | |
| | 10.3.3. | Reporting Standards for Pharmacokinetics | 24 |
| 10.4. | Appendi | x 4: Derived and Transformed Data | |
| | 10.4.1. | General | |
| | 10.4.2. | Study Population | 26 |
| | 10.4.3. | Safety | |
| 10.5. | Appendi | x 5: Reporting Standards for Missing Data | |
| | 10.5.1. | | |
| | 10.5.2. | Handling of Missing Data | |
| | | 10.5.2.1. Handling of Missing and Partial Dates | |
| 10.6. | Appendi | x 6: Division of AIDS (DAIDS) Table for Grading the | |
| | | of Adult and Pediatric Adverse Events | 29 |
| | 10.6.1. | Laboratory Values | |
| 10.7. | Appendi | x 7: Values of Potential Clinical Importance | |
| | | ECG | |
| | 10.7.2. | | |
| 10.8. | Appendi | x 8: Abbreviations & Trade Marks | |
| | 10.8.1. | Abbreviations | |
| | 10.8.2. | Trademarks | 33 |
| 10.9. | Appendi | x 9: List of Data Displays | 34 |
| | 10.9.1. | Data Display Numbering | 34 |
| | 10.9.2. | Mock Example Shell Referencing | |
| | 10.9.3. | Deliverables | |
| | 10.9.4. | Study Population Tables | 35 |
| | 10.9.5. | Safety Tables | |
| | 10.9.6. | Safety Figures | |
| | 10.9.7. | Pharmacokinetic Tables | |
| | 10.9.8. | Pharmacokinetic Figures | |
| | 10.9.9. | ICH Listings | |
| | 10.9.10. | • | |
| | | <b>-</b> | |

### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol: 208134

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

This is an open-label, single-sequence, one-way drug interaction study to investigate the effect of GSK3640254 on the pharmacokinetics (PK) of tenofovir alafenamide (TAF) and emtricitabine (FTC). Treatment of human immunodeficiency virus (HIV) infection frequently involves combination therapy. It is important to understand any interactions and resulting changes in exposure (if any) when HIV medications are given in combination. Data from this study will contribute to dosing recommendations when GSK3640254 and TAF/FTC are given in combination.

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol (Dated: 27/DEC/2018).

# 2.2. Study Objective(s) and Endpoint(s)

| Ob | jectives | En | dpoints |
|---|---|---|---|
| Pri | imary Objectives | Pri | Primary Endpoints |
| • | To assess the effect of GSK3640254 on the PK of TAF, FTC, and the active metabolite of TAF prodrug, TFV under fed conditions in healthy participants | • | AUC from Time 0 to the End of the Dosing Interval at Steady State (AUC(0- $\tau$ )) and Maximum Observed Concentration (Cmax) for TAF AUC(0- $\tau$ ), Cmax, and C $\tau$ for FTC and TFV |
| Se | condary Objectives | Se | condary Endpoints |
| • | To assess the safety and tolerability of TAF/FTC administered alone and when coadministered with GSK3640254 in healthy participants | • | Safety and tolerability parameters for Adverse Events (AEs)/Serious Adverse Events (SAEs), observed and change from baseline clinical laboratory assessments, electrocardiograms (ECGs), and vital sign measurements |
| • | To characterize the steady-state PK of GSK3640254 in the presence of TAF/FTC in healthy participants | • | AUC(0- $\tau$ ), Cmax, C $\tau$ , and Time of Maximum Observed Concentration (Tmax) for GSK3640254 |
| • | To characterize the steady-state PK of TAF, FTC, and TFV alone and in combination with GSK3640254 in healthy participants | • | Tmax for TAF, FTC, and TFV |

# 2.3. Study Design



# 2.4. Statistical Hypotheses

No formal research hypothesis that will be statistically tested in this study.

Coadministration of GSK3640254 and TAF and FTC may increase the exposure of TAF, FTC, and the metabolite TFV, and coadministration of GSK3640254 with TAF and FTC are expected to have no significant impact on the exposure of GSK3640254.

Analyses will be performed on the natural logarithms of AUC(0- $\tau$ ), C $\tau$  and Cmax using linear mixed-effect models with period as a fixed effect, participants as random effect, and measurements within participant as repeated measures. Effects will be estimated, and confidence intervals (CIs) will be constructed for the following treatment comparisons:

• Period 2 versus Period 1 (TAF, FTC, and TFV)

# 3. PLANNED ANALYSES

# 3.1. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who signed the informed consent form | Study Population |
| Safety | <ul> <li>All participants who received at least 1 dose of study medication.</li> <li>This population will be used for all demographic and safety summaries</li> </ul> | <ul><li>Study Population</li><li>Safety</li></ul> |
| Pharmacokinetic<br>Concentration | <ul> <li>All participants who underwent plasma PK sampling and had evaluable PK assay results.</li> <li>This population will be used for the PK concentration listings, summary tables, and plotting of concentration-time data.</li> </ul> | PK Concentration |
| Pharmacokinetic<br>Parameter | <ul> <li>All participants who underwent plasma PK sampling and had evaluable PK parameters estimated.</li> <li>This population will be used for PK parameter listings, summary tables, and statistical analysis tables.</li> </ul> | <ul><li>PK Parameter</li><li>PK statistical<br/>analysis</li></ul> |

Refer to Appendix 9: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, participant management or participant assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan dated 11MAR2019. The "significant" protocol deviation in the Protocol Deviation Management Plan is equivalent to "important" protocol deviations.

- Data will be reviewed prior to freezing the database to ensure all significant deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate listing of all inclusion/exclusion criteria deviations will also be provided. This listing will be based on data as recorded on the inclusion/exclusion page of the electronic case record form (eCRF).

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | |
|---|---|---|
| Data Displays for Reporting | | |
| Description Code Order in TLF | | |
| TAF/FTC 25/200 mg QD on Days 1 through 14 in Period 1 | TAF/FTC | 1 |
| TAF/FTC 25/200 mg QD + GSK3640254 200 mg QD on Days 1 through 7 in Period 2 | TAF/FTC+GSK3640254 | 2 |

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions), the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline. Baseline is applied to each treatment period.

| Parameter | Study As | sessment<br>Basel | s Considered as<br>ine | Baseline Used in Data Displa | |
|---|---|---|---|---|---|
| | Screening | Day -1 | Day 1 (Pre-Dose) | Period 1 Period 2 | |
| Safety | | | | | |
| Vital Sign | Х | Х | X | Day 1 (Pre-Dose) for each period | |
| 12-Lead ECG | Х | Χ | X | Day 1 (Pre-Dose)[1] for each period | |
| Hematology | Х | Χ | | Day -1 Period 1 Day 14 | |
| Clinical<br>Chemistry | Х | Х | | Day -1 Period 1 Day 1 | |
| Urinalysis | Х | Χ | | Day -1 | Period 1 Day 14 |

<sup>[1]</sup> The average (for quantitative assessments) or the worst case (for interpretation) of the predose triplicate assessments on Day 1 of Period 1 will be used as the baseline for Period 1. The average (for quantitative assessments) or the worst case (for interpretation) of the predose triplicate assessments on Day 1 of Period 2 will be used as the baseline for Period 2.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

# 5.3. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Schedule of Activities |
| 10.2 | Appendix 2: Study Phases and Treatment Emergent Adverse Events |
| 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| 10.4 | Appendix 4: Derived and Transformed Data |
| 10.5 | Appendix 5: Reporting Standards for Missing Data |
| 10.6 | Appendix 6: Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events |
| 10.7 | Appendix 7: Values of Potential Clinical Importance |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the "Safety" population, unless otherwise specified.

Study population analyses including analyses of participant's disposition, protocol deviations (including inclusion/exclusion criteria deviations), demographic and baseline characteristics, prior and concomitant medications, and exposure will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 9: List of Data Displays.

# 7. PHARMACOKINETIC ANALYSES

# 7.1. Primary Pharmacokinetic Analyses

#### 7.1.1. Endpoint / Variables

#### 7.1.1.1. Drug Concentration Measures

Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Standards for Pharmacokinetic). Plasma concentrations of GSK3640254, TAF, FTC, and TFV will be measured and reported.

#### 7.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin (6.4 or higher). All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| Сτ | Plasma concentration at the end of the dosing interval |
| AUC(0-τ) | Area under the plasma concentration-time curve from time 0 to the end of the dosing interval at steady state, to be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |

#### NOTES:

Additional parameters may be included as required.

#### 7.1.2. Summary Measure

Area under concentration-time curve (AUC(0- $\tau$ )), C $\tau$  and Cmax at steady state following doses of TAF/FTC 25/200 mg QD Days 1 through 14 in Period 1 and TAF/FTC 25/200 mg QD coadministered with GSK3640254 200 mg QD on Days 1 through 7 in Period 2 in healthy subjects.

#### 7.1.3. Population of Interest

The primary pharmacokinetic analyses will be based on the PK concentration population for plasma PK concentrations and the PK parameter population for plasma PK parameters and statistical analysis.

# 7.1.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

Primary plasma PK parameters (AUC(0- $\tau$ ) and Cmax) will be estimated for TAF (Periods 1 and 2) and primary plasma PK parameters AUC(0- $\tau$ ), C $\tau$ , and Cmax will be estimated for FTC and TFV (Periods 1 and 2). Summary statistics (arithmetic mean, geometric mean, median, standard deviation, minimum, maximum, and coefficient of variation) for plasma TAF, FTC, and TFV PK parameter values will be summarized by treatment

#### 7.1.4.1. Statistical Methodology Specification

The following PK statistical analyses will only be performed if sufficient data are available (i.e. if participants have well defined plasma profiles).

#### **Endpoint / Variables**

Plasma primary PK endpoints include AUC(0-τ), Cτ and Cmax, as data permit

#### **Model Specification**

- Analyses will be performed on the natural logarithms of AUC(0-τ), Cτ and Cmax using linear mixed-effect models with period as a fixed effect, participants as random effect, and measurements within participant as repeated measures.
- Effects will be estimated, and CIs will be constructed for the following treatment comparisons: Period 2 versus Period 1 (TAF, FTC, and TFV)
- Point estimates and 90% CIs for treatment differences on the log scale derived from the model will be exponentiated to obtain estimates for geometric mean ratios and CIs on the original scale.

### **Model Checking & Diagnostics**

 Model assumptions will be applied, but appropriate adjustments may be made based on the data.

#### **Model Results Presentation**

 Statistical analysis by analysis of variance (ANOVA) will be presented in tabular format with geometric mean ratios for:

Period 2 versus Period 1 (TAF, FTC, and TFV)

# 7.2. Secondary Pharmacokinetic Analyses

#### 7.2.1. Endpoint / Variables

#### 7.2.1.1. Drug Concentration Measures

Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Standards for Pharmacokinetic).

#### 7.2.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin (6.4 or higher). All calculations of non-compartmental parameters will be based on actual sampling times.

Plasma pharmacokinetic parameters listed below will be determined from the total plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. (GSK3640254 only) |
| Сτ | Plasma concentration at the end of the dosing interval (GSK3640254 only) |
| AUC(0-τ) | Area under the plasma concentration-time curve from time 0 to the end of the dosing interval at steady state, to be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. (GSK3640254 only) |
| Tmax | Time to first occurrence of Cmax |

#### NOTES:

Additional parameters may be included as required.

# 7.2.2. Summary Measure

Area under concentration-time curve [AUC(0- $\tau$ )], C $\tau$ , Cmax, and Tmax at steady state following doses of TAF/FTC 25/200 mg QD Days 1 through 14 in Period 1 and TAF/FTC 25/200 mg QD coadministered with GSK3640254 200 mg QD on Days 1 through 7 in Period 2 in healthy subjects.

#### 7.2.3. Population of Interest

The secondary pharmacokinetic analyses will be based on the PK concentration population for plasma PK concentrations, and the PK parameter population for plasma and statistical analysis, unless otherwise specified.

#### 7.2.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints/variables defined in Section 7.2.1 will be summarized using descriptive statistics, graphically presented (where appropriate) and listed.

Secondary plasma PK parameters (Tmax) will be estimated for TAF, FTC, and TFV (Periods 1 and 2) and secondary plasma PK parameters AUC(0- $\tau$ ), C $\tau$ , Cmax, and Tmax will be estimated for GSK3640254 (Period 2). Summary statistics (arithmetic mean, geometric mean, median, standard deviation, minimum, maximum, and coefficient of variation) for plasma GSK3640254 and TAF, FTC, and TFV PK parameter values will be summarized by treatment.

Predose (trough) PK plasma concentrations (TAF, FTC, and TFV: Days 2 through 14 [Period 1] and Days 1 through 7 [Period 2]; GSK3640254: Days 2 through 7 [Period 2]) will be summarized using the PK Concentration Population, and used to assess achievement of steady state.

# 8. SAFETY ANALYSES

The safety analyses will be based on the "Safety" population, unless otherwise specified.

### 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of AEs, SAEs and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 9: List of Data Displays.

# 8.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of chemistry laboratory tests, hematology laboratory tests, urinalysis, and liver function tests will be based on GSK Core Data Standards and will be graded using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (Version 2.1, July 2017). The details of the planned displays are in Appendix 9: List of Data Displays.

# 8.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs, vital signs, and Columbia Suicide Severity Rating Scale (C-SSRS) will be based on GSK Core Data Standards, unless otherwise specified. A figure of mean change from baseline in QTcF interval along with the 2-sided 95% CI using Student's t distribution will be presented by treatment and visit. The details of the planned displays are presented in Appendix 9: List of Data Displays.

# 9. REFERENCES

ViiV Healthcare group of companies Document Number 2018N383314\_00 (27-DEC-2018): An Open-Label One-way Interaction Clinical Trial to Evaluate the Pharmacokinetic Interactions Between GSK3640254 and Tenofovir Alafenamide/Emtricitabine in Healthy Subjects

# 10. APPENDICES

# 10.1. Appendix 1: Schedule of Activities

### 10.1.1. Protocol Defined Schedule of Events

# **Screening Visit**

| Procedure | Screening (up to 28 days before Day 1) |
|---|---|
| Outpatient visit | Χ |
| Informed consent | Х |
| Inclusion and exclusion criteria | Х |
| Demography | Х |
| Full physical examination including height and weight <sup>1</sup> | Х |
| Laboratory assessments (hematology, chemistry, urinalysis) | Х |
| 12-lead electrocardiogram | Х |
| Vital sign measurements | Х |
| Medication/drug/alcohol history | Х |
| Past and current medical conditions | Х |
| Columbia Suicide Severity Rating Scale | Х |
| Serum pregnancy test | Х |
| Follicle-stimulating hormone (as needed, to confirm postmenopausal status) | Χ |
| Drug, alcohol, and cotinine screen | Χ |
| HIV, Hepatitis B and C screening | Χ |

HIV = human immunodeficiency virus.

A full physical examination will include at a minimum, assessments of the skin, cardiovascular, respiratory, gastrointestinal, and neurological systems.

# **Time and Events Table**

| Period 1 | | Period 2 | | | | | | | | Follow-u | р | Notes | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Day<br>–1 | Day<br>1-5 | Day<br>6-13 | Day<br>14 | Day 1 | Day 2 | Day 3 | Day 4 | Day 5 | Day 6 | Day 7 | Day 8 | Day 9 <sup>1</sup> | Day 10 | |
| Admit to clinic | Х | | | | | | | | | | | | | | |
| Discharge from clinic | | | | | | | | | | | | | | Х | |
| Brief physical examination | X | | | | | | | | | | | | Х | | A brief physical examination will include, at a minimum, assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen). |
| Vital sign measurements | Χ | Χ | D7 | | Χ | | | Χ | | | Χ | | Χ | Х | |
| Single 12-lead ECG | Х | D1 | | | X | | | X | | | X | | X | | All ECGs in Period 1<br>and 2 will be pre-dose,<br>post-dose at 2 hours,<br>and post-dose 4 hours.<br>The predose ECGs on<br>Day 1 of both Period 1<br>and Period 2 will be<br>taken in triplicate. |
| Drug, alcohol, and cotinine screen | Х | | | | | | | | | | | | | | See Protocol Appendix 2 for specific tests to be performed. |
| Laboratory assessments (hematology, chemistry, urinalysis) | Х | | D7 | Х | | | Х | | | | Х | | Х | | See Protocol Appendix 2 for specific tests to be performed. |
| Pregnancy test | Χ | | | | | | | | | | | | Χ | | |
| Columbia-Suicide Severity<br>Rating Scale | | | | | Х | | | | | | Х | | | | |

| | Period 1 | | | | Period 2 | | | | | | | | Follow-u | p | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Day<br>-1 | Day<br>1-5 | Day<br>6-13 | Day<br>14 | Day 1 | Day 2 | Day 3 | Day 4 | Day 5 | Day 6 | Day 7 | Day 8 | Day 9 <sup>1</sup> | Day 10 | |
| Genetic sample (Optional) | Х | | | | | | | | | | | | | | |
| Study intervention:<br>TAF/FTC 25/200 mg | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | | | |
| Study intervention:<br>GSK3640254 200 mg | | | | | Х | Х | Х | Х | Х | Х | Х | | | | |
| TAF, FTC, and TFV serial<br>PK sampling | | | | х | х | | | | | | х | Х | | | Blood collection for PK analysis of TAF, FTC, and TFV will be collected at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours postdose (Period 1, Day 14 and Period 2, Day 7). |
| TAF, FTC, and TFV trough PK sampling | | D2-5 | Х | Х | Х | Х | Х | Х | Х | Х | Х | | | | Blood collection for TAF,<br>FTC, and TFV trough<br>PK samples will be<br>collected on Period 1,<br>Days 2 through 14 and<br>Period 2, Days 1<br>through 7. |
| GSK3640254 serial PK sampling | | | | | | | | | | | Х | Х | | | Blood collection for PK analysis of GSK3640254 will be collected at 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, and 24 hours postdose (Period 2, Day 7). |

| | Period 1 | | | | Period 2 | | | | | | | | р | Notes | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Day<br>–1 | Day<br>1-5 | Day<br>6-13 | Day<br>14 | Day 1 | Day 2 | Day 3 | Day 4 | Day 5 | Day 6 | Day 7 | Day 8 | Day 91 | Day 10 | |
| GSK3640254 trough PK sampling | | | | | | Х | Х | Х | Х | Х | Х | | | | Blood collection for<br>GSK3640254 trough PK<br>samples will be<br>collected on Period 2,<br>Days 2 through 7. |
| AE review | | ←=====→ | | | | | | | | | | | | | |
| SAE review | ←======→ | | | | | | | | | | | | | | |
| Concomitant medication review | + | ===== | | | ====== | ===== | ====== | ===== | ===== | ===== | ===== | ===== | ====== | ==-> | |

AE = adverse event; D = Day; ECG = electrocardiogram; FTC = emtricitabine; PK = pharmacokinetic; SAE = serious adverse event; TAF = tenofovir alafenamide; TFV = tenofovir; W = washout.

<sup>1</sup> Evaluations scheduled for Period 2, Day 9 will also be performed for participants who discontinue early.

# 10.2. Appendix 2: Study Phases and Treatment Emergent Adverse Events

# 10.2.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment start date(/time) and stop date(/time).

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date and Time ≤ Study Treatment Start Date and Time |
| On-Treatment | Study Treatment Start Date and Time < Date and Time ≤ Study Treatment Stop Date and Time + 4 days |
| Post-Treatment | Date and Time > Study Treatment Stop Date and Time + 4 days |

### 10.2.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before Day -1 of Period 1 |
| Concomitant | Any medication that is not a prior |

#### NOTES:

• Please refer to Appendix 5: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 10.2.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | <ul> <li>If AE onset date and time is on or after treatment start date and time &amp; on or before treatment stop date and time + 4 days.</li> <li>Study Treatment Start Date and Time ≤ AE Start Date and Time ≤ Study Treatment Stop Date and Time + 4 days.</li> <li>If the AE onset date is completely missing, the AE is considered as treatment emergent.</li> </ul> |

### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Please refer to Appendix 5: Reporting Standards for Missing Data for handling of missing and partial dates for adverse events. Use the rules in this table if the adverse event onset date is completely missing.

# 10.3. Appendix 3: Data Display Standards & Handling Conventions

# 10.3.1. Reporting Process

| Software | |
|---|---|
| The currently support the currently support to the currently suppo | The currently supported versions of SAS software (9.4 or higher) will be used. |
| Reporting Area | Reporting Area |
| HARP Server | Not applicable |
| HARP Compound Not applicable | |
| Analysis Datasets | |

- Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 & ADaM IG Version 1.1).
- For creation of ADaM datasets (ADC1/ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### **Generation of RTF Files**

RTF files will be generated for all reporting efforts described in the RAP.

### 10.3.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include participant level listings in the main body of the GSK Clinical Study Report. All
  participant level listings should be located in the modular appendices as ICH or non-ICH listings.

#### **Formats**

- All data will be reported according to the actual treatment the participant received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures, and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the participant's listings.

• Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures (mean figures only for PK concentrations), summaries and statistical analyses (excluding statistical analyses of PK parameters).

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables except for determining the worst-case values.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

# 10.3.3. Reporting Standards for Pharmacokinetics

| DI LI CIO | D |
|---|---|
| Pharmacokinetic Con | |
| Descriptive Summary | Refer to IDSL PK Display Standards. |
| Statistics, Graphical | Refer to IDSL Statistical Principle 6.06.1. |
| Displays and Listings | For continuous data: |
| | <ul> <li>NQs at the beginning of a participant profile (i.e. before the first incidence of a measurable concentration) are deemed to be zero as it is assumed that in this circumstance no drug is yet measurable in the blood.</li> <li>For NQs at the end of the participant profile (i.e. after the last incidence of a measurable concentration);</li> <li>for individual plots and pharmacokinetic analyses these are dropped (set to missing) as they do not provide any useful information (and can erroneously indicate that absolutely no drug is present)</li> <li>for summary statistics, these are set to 0 (to avoid skewing of the summary statistics)</li> <li>Individual NQs which fall between two measurable concentrations are set to missing (individual values of this nature are assumed to be an anomaly)</li> <li>If two or more NQ values occur in succession between measurable concentrations, the profile will be deemed to have terminated at the last measurable concentration prior to these NQs. For the purpose of individual participant plots, these NQs will be set to 0, and the subsequent measurable concentrations will be retained. For the derivation of pharmacokinetic parameters, these NQs and any subsequent measurable concentrations will be omitted (set to missing).</li> </ul> |
| | Note: Concentration values will be imputed as per GUI_51487 for descriptive |
| | summary statistics/analysis and summarized graphical displays only. |
| Pharmacokinetic Para | ameter Data |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | N, n, geometric mean, 95% CI of geometric mean, SD of logged data and between-<br>subject geometric coefficient of variation (CVb (%)) will be reported.<br>CV <sub>b</sub> (%) = √ (exp(SD²) - 1) * 100<br>(SD = SD of Ln-Transformed data) |
| Parameters Not<br>Being Ln-<br>Transformed | Tmax, λz, λz lower, λz upper, and λz no. of points. |

| Parameters Not<br>Being Summarized | λz, λz lower, λz upper, and λz no. of points. |
|---|---|
| Listings | Include the first point, last point and number of points used in the determination of λz and Rsq_adjusted for listings. |

# 10.4. Appendix 4: Derived and Transformed Data

#### 10.4.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- The worst finding/interpretation associated with multiple measurements as the finding/interpretation for that time point.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from First Dose Date in Period 1:
  - Assessment Date = Missing → Study Day = Missing
  - Assessment Date < First Dose Date in Period 1 → Study Day = Assessment Date First Dose
    Date</li>
  - Assessment Date >= First Dose Date in Period 1 → Study Day = Assessment Date (First Dose Date in Period 1) + 1

#### **Period Day**

- Calculated as the number of days from First Dose Date for the respective period:
  - Assessment Date = Missing 
    → Study Day = Missing
  - Assessment Date < First Dose Date in Period 1 → Study Day = Assessment Date First Dose
    Date</li>
  - First Dose Date in Period 1 <= Assessment Date < First Dose Date in Period 2 → Study Day =
     Assessment Date (First Dose Date in Period 1) + 1</li>
  - Assessment Date >= First Dose Date in Period 2 → Study Day = Assessment Date (First Dose Date in Period 2) + 1

# 10.4.2. Study Population

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any participant with a missing day will have this imputed as day '15'.
  - Any participant with a missing day and month will have this imputed as PPD
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

# 10.4.3. Safety

# Adverse Events

# **AEs of Special Interest**

No analysis for AEs of Special Interest will be performed

# 10.5. Appendix 5: Reporting Standards for Missing Data

# 10.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Participant study completion (i.e. as specified in the protocol) was defined as the participant has completed all phases of the study including the final date on which data were or are expected to be collected.</li> <li>Withdrawn participants were not replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 10.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in participant listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 10.5.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in participant listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 2: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied.</li> </ul> |
| | Consequently, time to onset and duration of such events will be missing. |
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the eCRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | <ul> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 10.6. Appendix 6: Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events

# 10.6.1. Laboratory Values

Laboratory abnormalities will be graded according to the DAIDS grading table Version 2.1, July 2017. Laboratory results are converted to use SI units; only the numeric part of the criteria will be used. If for a laboratory parameter there are multiple grades sharing the same criteria, the maximum grade will be used.

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Absolute Lymphocyte Count, Low (cell/mm³; cells/L) > 5 years of age (not HIV infected) | 600 to < 650<br>0.600 × 10 <sup>9</sup> to < 0.650 × 10 <sup>9</sup> | 500 to < 600<br>0.500 × 10 <sup>9</sup> to < 0.600 ×<br>10 <sup>9</sup> | 350 to < 500<br>0.350 × 10 <sup>9</sup> to < 0.500 × 10 <sup>9</sup> | < 350<br>< 0.350 × 10 <sup>9</sup> |
| Absolute Neutrophil Count, Low (cells/mm³; cells/L) > 7 days of age | 800 to 1,000<br>0.800 × 10 <sup>9</sup> to 1.000 × 10 <sup>9</sup> | 600 to 799<br>0.600 × 10 <sup>9</sup> to 0.799 ×<br>10 <sup>9</sup> | 400 to 599<br>0.400 × 10 <sup>9</sup> to 0.599 × 10 <sup>9</sup> | < 400<br>< 0.400 × 10 <sup>9</sup> |
| Hemoglobin, Low (g/dL; mmol/L) | 10.0 to 10.9 | 9.0 to < 10.0 | 7.0 to < 9.0 | < 7.0 |
| ≥ 13 years of age (male only) | 6.19 to 6.76 | 5.57 to < 6.19 | 4.34 to < 5.57 | <4.34 |
| Hemoglobin, Low (g/dL; mmol/L) | 9.5 to 10.4 | 8.5 to < 9.5 | 6.5 to < 8.5 | < 6.5 |
| ≥ 13 years of age (female only) | 5.88 to 6.48 | 5.25 to < 5.88 | 4.03 to < 5.25 | < 4.03 |
| Platelets, Decreased (cells/mm³; cells/L) | 100,000 to < 125,000<br>100.000 × 10 <sup>9</sup> to < 125.000<br>× 10 <sup>9</sup> | 50,000 to < 100,000<br>50.000 × 10 <sup>9</sup> to <<br>100.000 × 10 <sup>9</sup> | 25,000 to < 50,000<br>25.000 × 10 <sup>9</sup> to < 50.000 ×<br>10 <sup>9</sup> | < 25,000<br>< 25.000 × 10 <sup>9</sup> |
| White Blood Cell, Decreased (cells/mm³; cells/L) > 7 days of age | 2,000 to 2,499<br>2.000 × 10 <sup>9</sup> to 2.499 × 10 <sup>9</sup> | 1,500 to 1,999<br>1.500 × 10 <sup>9</sup> to 1.999 ×<br>10 <sup>9</sup> | 1,000 to 1,499<br>1.000 × 10 <sup>9</sup> to 1.499 × 10 <sup>9</sup> | < 1,000<br>< 1.000 × 10 <sup>9</sup> |

| Clinical Chemistry | | | | |
|--------------------------|--------------|----------------|---------|---------|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Albumin Low (ald : all ) | 3.0 to < LLN | ≥ 2.0 to < 3.0 | < 2.0 | NA |
| Albumin, Low (g/dL; g/L) | 30 to < LLN | ≥ 20 to < 30 | < 20 | NA |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Alkaline Phosphatase, High | 1.25 to < 2.5 × ULN | 2.5 to < 5.0 × ULN | 5.0 to < 10.0 × ULN | ≥ 10.0 × ULN |
| Alanine Aminotransferase, High | 1.25 to < 2.5 × ULN | 2.5 to < 5.0 × ULN | 5.0 to < 10.0 × ULN | ≥ 10.0 ULN |
| Amylase (Total), High | 1.1 to < 1.5 × ULN | 1.5 to < 3.0 × ULN | 3.0 to < 5.0 × ULN | ≥ 5.0 × ULN |
| Aspartate Aminotransferase, High | 1.25 to < 2.5 × ULN | 2.5 to < 5.0 × ULN | 5.0 to < 10.0 × ULN | ≥ 10.0 × ULN |
| Bicarbonate, Low (mEq/L; mmol/L) | 16.0 to < LLN<br>16.0 to < LLN | 11.0 to < 16.0<br>11.0 to < 16.0 | 8.0 to < 11.0<br>8.0 to < 110. | < 8.0<br>< 8.0 |
| Direct Bilirubin, High > 28 days of age | NA | NA | > ULN with other signs and symptoms of hepatotoxicity | > ULN with life-threatening consequences (e.g., signs and symptoms of liver failure) |
| Total Bilirubin, High > 28 days of age | 1.1 to < 1.6 × ULN | 1.6 to < 2.6 × ULN | 2.6 to < 5.0 × ULN | ≥ 5.0 × ULN |
| Calcium, High (mg/dL; mmol/L) | 10.6 to < 11.5 | 11.5 to < 12.5 | 12.5 to < 13.5 | ≥ 13.5 |
| ≥ 7 days of age | 2.65 to < 2.88 | 2.88 to < 3.13 | 3.13 to < 3.38 | ≥ 3.38 |
| Calcium, Low (mg/dL; mmol/L) | 7.8 to < 8.4 | 7.0 to < 7.8 | 6.1 to < 7.0 | < 6.1 |
| ≥ 7 days of age | 1.95 to < 2.10 | 1.75 to < 1.95 | 1.53 to < 1.75 | < 1.53 |
| Creatine Kinase, High | 3 to < 6 × ULN | 6 to < 10 × ULN | 10 to < 20 × ULN | ≥ 20 × ULN |
| Creatinine, High Choose the method that selects for the higher grade | 1.1 to 1.3 × ULN | > 1.3 to 1.8 × ULN OR<br>Increase to 1.3 to < 1.5 ×<br>participant's baseline | > 1.8 to < 3.5 ULN OR<br>Increase to 1.5 to < 2.0 ×<br>participant's baseline | ≥ 3.5 × ULN OR Increase of ≥ 2.0 × participant's baseline |
| Glucose Fasting, High (mg/dL; mmol/L) | 110 to 125<br>6.11 to < 6.95 | > 125 to 250<br>6.95 to < 13.89 | > 250 to 500<br>13.89 to < 27.75 | ≥ 500<br>≥ 27.75 |
| Glucose, Low (mg/dL; mmol/L) ≥ 1 month of age | 55 to 64<br>3.05 to < 3.55 | 40 to < 55<br>2.22 to < 3.05 | 30 to < 40<br>1.67 to < 2.22 | < 30<br>< 1.67 |
| Lipase, High | 1.1 to < 1.5 × ULN | 1.5 to < 3.0 × ULN | 3.0 to < 5.0 × ULN | ≥ 5.0 × ULN |
| Cholesterol, Fasting, High (mg/dL;<br>mmol/L)<br>≥ 18 years of age | 200 to < 240<br>5.18 to < 6.19 | 240 to < 300<br>6.19 to < 7.77 | ≥ 300<br>≥ 7.77 | NA |
| Triglycerides, Fasting, High (mg/dL; mmol/L) | 150 to 300<br>1.71 to 3.42 | > 300 to 500<br>> 3.42 to 5.7 | > 500 to < 1.000<br>> 5.7 to 11.4 | > 1,000<br>> 11.4 |
| Phosphate, Low (mg/dL; mmol/L) > 14 years of age | 2.0 to < LLN<br>0.65 to < LLN | 1.4 to < 2.0<br>0.45 to < 0.65 | 1.0 to < 1.4<br>0.32 to < 0.45 | < 1.0<br>< 0.32 |
| Potassium, High (mEq/L; mmol/L) | 5.6 to < 6.0<br>5.6 to < 6.0 | 6.0 to < 6.5<br>6.0 to < 6.5 | 6.5 to < 7.0<br>6.5 to < 7.0 | ≥ 7.0<br>≥ 7.0 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Potossium Low (mEa/L: mmol/L) | 3.0 to < 3.4 | 2.5 to < 3.0 | 2.0 to < 2.5 | < 2.0 |
| Potassium, Low (mEq/L; mmol/L) | 3.0 to < 3.4 | 2.5 to < 3.0 | 2.0 to < 2.5 | < 2.0 |
| Codina High (mFa/L) | 146 to < 150 | 150 to < 154 | 154 to < 160 | ≥ 160 |
| Sodium, High (mEq/L; mmol/L) | 146 to < 150 | 150 to < 154 | 154 to < 160 | ≥ 160 |
| Codium Lourine Fall Lourine (III) | 130 to < 135 | 125 to < 130 | 121 to < 125 | ≤ 120 |
| Sodium, Low (mEq/L; mmol/L) | 130 to < 135 | 125 to < 130 | 121 to < 125 | ≤ 120 |
| Usia Asid High (mFa/L, mmal/L) | 7.5 to < 10.0 | 10.0 to < 12.0 | 12.0 to < 15.0 | ≥ 15.0 |
| Uric Acid, High (mEq/L; mmol/L) | 0.45 to < 0.59 | 0.59 to < 0.71 | 0.71 to < 0.89 | ≥ 0.89 |

NA=not applicable; LLN = lower limit of normal; ULN=upper limit of normal.

| Urinalysis | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Glucose/Glycosuria (random collection tested by dipstick) | Trace to 1+ or ≤ 250 mg | 2+ or > 250 to ≤ 500 mg | > 2+ or > 500 mg | NA |
| Protein/Proteinuria (random collection tested by dipstick) | 1+ | 2+ | 3+ or higher | NA |
| Red Blood Cells (RBCs)/Hematuria (not<br>to be reported based on dipstick findings<br>or on blood believed to be of menstrual<br>origin) | 6 to < 10 RBCs per high<br>power field | ≥ 10 RBCs per high power field | Gross, with or without clots<br>OR with RBC casts OR<br>intervention indicated | Life-threatening consequences |

NA=not applicable

# 10.7. Appendix 7: Values of Potential Clinical Importance

# 10.7.1. ECG

| ECG Parameter | Units | Potential Clinically | y Important Range |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | <320 | >450 |
| Absolute PR Interval | msec | < 120 | > 200 |
| Absolute QRS Interval | msec | < 60 | > 120 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | > 60 |

# 10.7.2. Vital Signs

| Vital Sign Parameter | Units | Potential Clinically Important Range | |
|---|---|---|---|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 140 |
| Diastolic Blood Pressure | mmHg | < 45 | > 90 |
| Heart Rate | bpm | < 40 | > 100 |

# 10.8. Appendix 8: Abbreviations & Trade Marks

# 10.8.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AUC | Area under the Plasma Concentration-Time Curve |
| AUC(0-τ) | AUC from Time 0 to the End of the Dosing Interval at Steady State |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| Cmax | Maximum Observed Concentration |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| Cτ | Plasma Concentration at the End of the Dosing Interval |
| CV <sub>b</sub> | Coefficient of Variation (Between) |
| DBF | Database Freeze |
| DBR | Database Release |
| DP | Decimal Places |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| FTC | Emtricitabine |
| GSK | GlaxoSmithKline |
| HIV | human immunodeficiency virus |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| LLN | Lower Limit of Normal |
| PK | Pharmacokinetic |
| QD | Once Daily |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SD | Standard Deviation |
| SDTM | Study Data Tabulation Model |
| TAF | Tenofovir Alafenamide |
| TFV | Tenofovir |
| Tmax | Time of Maximum Observed Concentration |
| ULN | Upper Limit of Normal |

# 10.8.2. Trademarks

| Trademarks of the GlaxoSmit<br>Group of Companies | hKline |
|---------------------------------------------------|--------|
| NONE | |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |
| WinNonlin |

# 10.9. Appendix 9: List of Data Displays

# 10.9.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|-------------|
| Study Population | 1.1 to 1.7 | |
| Safety | 2.1 to 2.19 | 2.1 |
| Pharmacokinetic | 3.1 to 3.19 | 3.1 to 3.20 |
| Section | Listings | |
| ICH Listings | 1 to 30 | |
| Other Listings | 31 to 37 | |

# 10.9.2. Mock Example Shell Referencing

Non-IDSL specifications will be referenced as indicated and if required example mock-up displays provided in the Table/Listing/Figure Shells.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

#### NOTES:

• Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 10.9.3. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

# 10.9.4. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | Safety | NS1 | Summary of Number of Subjects Enrolled by Country and Site ID | | SAC |
| 1.2. | Safety | ES1A | Summary of Subject Disposition for the Subject Conclusion Record | | SAC |
| 1.3. | Screened | SD1 | Summary of Screening Status and Reasons for Screen Failures | | SAC |
| Protoc | ol Deviation | | | | |
| 1.4. | Safety | DV1 | Summary of Important Protocol Deviations | | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.5. | Safety | DM3 | Summary of Demographic Characteristics | | SAC |
| 1.6. | Safety | DM5 | Summary of Race and Racial Combinations | | SAC |
| 1.7. | Safety | DM11 | Summary of Age Ranges | | SAC |

# 10.9.5. Safety Tables

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | • | |
| 2.1. | Safety | AE1CP | Summary of Adverse Events by System Organ Class and Preferred Term | | SAC |
| 2.2. | Safety | AE1CP | Summary of Drug-Related Adverse Events by System Organ Class and Preferred Term | | SAC |
| 2.3. | Safety | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency | | SAC |
| 2.4. | Safety | AE15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC |
| 2.5. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC |
| 2.6. | Safety | AE5A | Summary of Adverse Events by System Organ Class and Preferred Term and Maximum Intensity | | SAC |
| Labora | tory: Chemistry | / | | | • |
| 2.7. | Safety | LB1 | Summary of Clinical Chemistry Changes from Baseline | | SAC |
| 2.8. | Safety | LB16 | Summary of Clinical Chemistry Results by Maximum Grade Increase Post-Baseline Relative to Baseline | | SAC |
| Labora | tory: Hematolo | gy | | • | |
| 2.9. | Safety | LB1 | Summary of Hematology Changes from Baseline | | SAC |
| 2.10. | Safety | LB16 | Summary of Hematology Results by Maximum Grade Increase Post-Baseline Relative to Baseline | | SAC |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory: Urinalysis | ; | | | |
| 2.11. | Safety | UR3 | Summary of Urinalysis Dipstick Results | | SAC |
| 2.12. | Safety | LB1 | Summary of Urine Concentration Changes from Baseline | | SAC |
| 2.13. | Safety | LB16 | Summary of Urinalysis by Maximum Grade Increase Post-<br>Baseline Relative to Baseline | | SAC |
| ECG | | | | | |
| 2.14. | Safety | EG1 | Summary of ECG Findings | | SAC |
| 2.15. | Safety | EG2 | Summary of ECG Changes from Baseline | | SAC |
| 2.16. | Safety | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category | | SAC |
| 2.17. | Safety | EG11 | Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category | | SAC |
| Vital Si | gns | | | | |
| 2.18. | Safety | VS1 | Summary of Vital Sign Changes from Baseline | | SAC |
| C-SSR | S | | | | |
| 2.19. | Safety | CSSRS4 | Listing of C-SSRS Suicidal Ideation and Behavior Data | Only include participants who have suicidal ideation or behavior | SAC |

# 10.9.6. Safety Figures

| Safety: | Safety: Tables | | | |
|---|---|---|---|---|
| No. | o. Population IDSL / Example Shell Title Programming Notes Deliverab [Priority] | | | |
| ECG | | | | |
| 2.1. | Safety | EG9 | Mean (95% CI) Change from Baseline in QTcF Interval by Timepoint and Treatment | SAC |

# 10.9.7. Pharmacokinetic Tables

| Pharm | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Concentration Data | | | | | |
| 3.1. | PK<br>Concentration | PKCT1 | Summary of Tenofovir Alafenamide (TAF) Plasma Pharmacokinetic Concentration-Time Data (units) by Treatment | | SAC |
| 3.2. | PK<br>Concentration | PKCT1 | Summary of Tenofovir (TFV) Plasma Pharmacokinetic Concentration-Time Data (units) by Treatment | | SAC |
| 3.3. | PK<br>Concentration | PKCT1 | Summary of Emtricitabine (FTC) Plasma Pharmacokinetic Concentration-Time Data (units) by Treatment | | SAC |
| 3.4. | PK<br>Concentration | PKCT1 | Summary of GSK3640254 Plasma Pharmacokinetic Concentration-Time Data (units) by Treatment | | SAC |
| 3.5. | PK<br>Concentration | PKCT1 | Summary of Predose (trough) Tenofovir Alafenamide (TAF) Plasma Concentration Data (units) by Treatment | | SAC |
| 3.6. | PK<br>Concentration | PKCT1 | Summary of Predose (trough) Tenofovir (TFV) Plasma<br>Concentration Data (units) by Treatment | | SAC |
| 3.7. | PK<br>Concentration | PKCT1 | Summary of Predose (trough) Emtricitabine (FTC) Plasma Concentration Data (units) by Treatment | | SAC |
| 3.8. | PK<br>Concentration | PKCT1 | Summary of Predose (trough) GSK3640254 Plasma<br>Concentration Data (units) by Treatment | | SAC |
| PK Dei | rived Parameters | 3 | | | |
| 3.9. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived Tenofovir Alafenamide (TAF) Plasma Pharmacokinetic Parameters (Non-Transformed) Based on Actual Time by Treatment | Parameters with units | SAC |
| 3.10. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived Tenofovir Alafenamide (TAF) Plasma Pharmacokinetic Parameters (Ln-Transformed) Based on Actual Time by Treatment | Parameters with units | SAC |

| Pharma | acokinetic: Tabl | es | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.11. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived Tenofovir (TFV) Plasma Pharmacokinetic Parameters (Non-Transformed) Based on Actual Time by Treatment | Parameters with units | SAC |
| 3.12. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived Tenofovir (TFV) Plasma Pharmacokinetic Parameters (Ln-Transformed) Based on Actual Time by Treatment | Parameters with units | SAC |
| 3.13. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived Emtricitabine (FTC) Plasma<br>Pharmacokinetic Parameters (Non-Transformed) Based on<br>Actual Time by Treatment | Parameters with units | SAC |
| 3.14. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived Emtricitabine (FTC) Plasma Pharmacokinetic Parameters (Ln-Transformed) Based on Actual Time by Treatment | Parameters with units | SAC |
| 3.15. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived GSK3640254 Plasma<br>Pharmacokinetic Parameters (Non-Transformed) Based on<br>Actual Time by Treatment | Parameters with units | SAC |
| 3.16. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived GSK3640254 Plasma<br>Pharmacokinetic Parameters (Ln-Transformed) Based on Actual<br>Time by Treatment | Parameters with units | SAC |
| PK Ana | lysis Tables | | | | |
| 3.17. | PK<br>Parameter | PKPT3 | Statistical Analysis of Tenofovir Alafenamide (TAF) Plasma<br>Pharmacokinetic Parameters: Analysis of Variance (ANOVA) | AUC(0-τ), Cτ, and Cmax | SAC |
| 3.18. | PK<br>Parameter | PKPT3 | Statistical Analysis of Tenofovir (TFV) Plasma Pharmacokinetic Parameters: Analysis of Variance (ANOVA) | AUC(0-τ), Cτ, and Cmax | SAC |
| 3.19. | PK<br>Parameter | PKPT3 | Statistical Analysis of Emtricitabine (FTC) Plasma Pharmacokinetic Parameters: Analysis of Variance (ANOVA) | AUC(0-τ), Cτ, and Cmax | SAC |

# 10.9.8. Pharmacokinetic Figures

| Pharm | acokinetic: Figu | res | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individ | ual Concentration | on Plots | | | • |
| 3.1. | PK<br>Concentration | PKCF1P | Individual Tenofovir Alafenamide (TAF) Plasma Concentration-<br>Time Plots by Participant (Linear and Semi-Logarithmic) | Paginate by Participant Dashed line represents the LLQ Periods Overlaid | SAC |
| 3.2. | PK<br>Concentration | PKCF1P | Individual Tenofovir (TFV) Plasma Concentration-Time Plots by Participant (Linear and Semi-Logarithmic) | Paginate by Participant Dashed line represents the LLQ Periods Overlaid | SAC |
| 3.3. | PK<br>Parameter | PKCF2 | Individual Emtricitabine (FTC) Plasma Concentration-Time Plots by Participant (Linear and Semi-Logarithmic) | Periods Overlaid | SAC |
| 3.4. | PK<br>Concentration | PKCF2 | Individual GSK3640254 Plasma Concentration-Time Plots by Participant (Linear and Semi-Logarithmic) | Periods Overlaid | SAC |
| 3.5. | PK<br>Parameter | PKCF2 | Individual Tenofovir Alafenamide (TAF) Plasma Concentration-<br>Time Plots by Treatment (Linear and Semi-Logarithmic) | Periods Overlaid | SAC |
| 3.6. | PK<br>Parameter | PKCF2 | Individual Tenofovir (TFV) Plasma Concentration-Time Plots by Treatment (Linear and Semi-Logarithmic) | Periods Overlaid | SAC |
| 3.7. | PK<br>Concentration | PKCF2 | Individual Emtricitabine (FTC) Plasma Concentration-Time Plots by Participant (Linear and Semi-Logarithmic) | Periods Overlaid | SAC |
| 3.8. | PK<br>Concentration | PKCF1P | Individual GSK3640254 Plasma Concentration-Time Plots by Treatment (Linear and Semi-Logarithmic) | Periods Overlaid | SAC |
| Mean / | Median Concen | tration Plots | | | |
| 3.9. | PK<br>Concentration | PKCF1P | Mean (± Standard Deviation) Tenofovir Alafenamide (TAF) Plasma Concentration-Time Plots by Treatment (Linear and Semi-Logarithmic) | Periods Overlaid | SAC |

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.10. | PK<br>Concentration | PKCF1P | Mean (± Standard Deviation) Tenofovir (TFV) Plasma<br>Concentration-Time Plots by Treatment (Linear and Semi-<br>Logarithmic) | Periods Overlaid | SAC |
| 3.11. | PK<br>Concentration | PKCF1P | Mean (± Standard Deviation) Emtricitabine (FTC) Plasma Concentration-Time Plots by Treatment (Linear and Semi-Logarithmic) | Periods Overlaid | SAC |
| 3.12. | PK<br>Concentration | PKCF2 | Mean (± Standard Deviation) GSK3640254 Plasma<br>Concentration-Time Plots by Treatment (Linear and Semi-<br>Logarithmic) | Periods Overlaid | SAC |
| 3.13. | PK<br>Concentration | PKCF3 | Median (Range) Tenofovir Alafenamide (TAF) Plasma<br>Concentration-Time Plots by Treatment (Linear and Semi-<br>Logarithmic) | Periods Overlaid | SAC |
| 3.14. | PK<br>Concentration | PKCF3 | Median (Range) Tenofovir (TFV) Plasma Concentration-Time Plots by Treatment (Linear and Semi-Logarithmic) | Periods Overlaid | SAC |
| 3.15. | PK<br>Concentration | PKCF3 | Median (Range) Emtricitabine (FTC) Plasma Concentration-<br>Time Plots by Treatment (Linear and Semi-Logarithmic) | Periods Overlaid | SAC |
| 3.16. | PK<br>Concentration | PKCF3 | Median (Range) GSK3640254 Plasma Concentration-Time Plots by Treatment (Linear and Semi-Logarithmic) | Periods Overlaid | SAC |
| 3.17. | PK<br>Concentration | PKCF3 | Mean (± Standard Deviation) Predose (Trough) Tenofovir<br>Alafenamide (TAF) Plasma Concentration Plots by Treatment<br>(Linear and Semi-Logarithmic) | Periods Overlaid | SAC |
| 3.18. | PK<br>Concentration | PKCF2 | Mean (± Standard Deviation) Predose (Trough) Tenofovir (TFV) Plasma Concentration Plots by Treatment (Linear and Semi-<br>Logarithmic) | Periods Overlaid | SAC |

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.19. | PK<br>Concentration | PKCF2 | Mean (± Standard Deviation) Predose (Trough) Emtricitabine (FTC) Plasma Concentration Plots by Treatment (Linear and Semi-Logarithmic) | Periods Overlaid | SAC |
| 3.20. | PK<br>Concentration | PKCF2 | Mean (± Standard Deviation) Predose (Trough) GSK3640254<br>Plasma Concentration Plots by Treatment (Linear and Semi-<br>Logarithmic) | Periods Overlaid | SAC |

# 10.9.9. ICH Listings

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | • | · |
| 1. | Safety | ES3 | Listing of Reasons for Study Withdrawal | | SAC |
| 2. | Screened | DS7 | Listing of Reasons for Screen Failure | | SAC |
| Protoc | ol Deviations | | | | · |
| 3. | Safety | DV2 | Listing of Important Protocol Deviations | | SAC |
| 4. | Safety | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC |
| Popula | tions Analysed | | | | <u>.</u> |
| 5. | Safety | SP3A | Listing of Subjects Excluded from Any Population | | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 6. | Safety | DM2 | Listing of Demographic Characteristics | | SAC |
| 7. | Safety | DM9 | Listing of Race | | SAC |
| Prior a | nd Concomitan | t Medications | | | · |
| 8. | Safety | CM5 | Listing of Concomitant Medications | Based on GSK Drug Dictionary | SAC |
| Exposi | ire and Treatmo | ent Compliance | | | · |
| 9. | Safety | EX4 | Listing of Exposure Data | | SAC |
| 10. | Safety | POP_L1 | Listing of Meal Data | | SAC |
| Advers | e Events | | | | |
| 11. | Safety | AE2 | Listing of Relationship Between System Organ Class and Verbatim Text | | SAC |
| 12. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 13. | Safety | AE9CP | Listing of All Adverse Events | | SAC |
| Serious | s and Other Sig | nificant Adverse | Events | | · |
| 14. | Safety | AE9CP | Listing of Study Drug Related Adverse Events | | SAC |
| 15. | Safety | AE9CP | Listing of Serious Adverse Events (Fatal & Non-Fatal) | | SAC |
| 16. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | | SAC |
| 17. | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study | | SAC |
| Hepato | biliary (Liver) | | | | |
| 18. | Safety | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping Events | | SAC |
| 19. | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events | | SAC |
| All Lab | oratory | | | | |
| 20. | Safety | LB5A | Listing of Clinical Chemistry with any Toxicities | | SAC |
| 21. | Safety | LB5A | Listing of All Clinical Chemistry Data for Subjects with any Toxicities | | SAC |
| 22. | Safety | LB5A | Listing of Hematology with any Toxicities | | SAC |
| 23. | Safety | LB5A | Listing of All Hematology Data for Subjects with any Toxicities | | SAC |
| 24. | Safety | LB5A | Listing of Urinalysis with any Toxicities | | SAC |
| 25. | Safety | LB5A | Listing of All Urinalysis Data for Subjects with any Toxicities | | SAC |
| ECG | | | | | |
| 26. | Safety | EG6 | Listing of All ECG Findings | | SAC |
| 27. | Safety | EG6 | Listing of All Abnormal ECG Findings | | SAC |
| 28. | Safety | EG4 | Listing of All ECG Values | | SAC |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital Signs | | | | | |
| 29. | Safety | VS5 | Listing of All Vital Signs of Potential Clinical Importance | | SAC |
| 30. | Safety | VS5 | Listing of All Vital Signs for Subjects with any Value of Potential Clinical Importance | | SAC |

# 10.9.10. Non-ICH Listings

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharmacokinetics | | | | | |
| 31. | PK<br>Concentration | PKCL1P | Listing of Tenofovir Alafenamide (TAF) and Tenofovir (TFV) Plasma Concentration-Time Data by Treatment | | SAC |
| 32. | PK<br>Concentration | PKCL1P | Listing of Emtricitabine (FTC) Plasma Concentration-Time Data by Treatment | | SAC |
| 33. | PK<br>Concentration | PKPL1P | Listing of GSK3640254 Plasma Concentration-Time Data by Treatment | | SAC |
| 34. | PK<br>Parameter | PKPL1P | Listing of Tenofovir Alafenamide (TAF) Plasma Pharmacokinetic Parameters Based on Actual Time by Treatment | | SAC |
| 35. | PK<br>Parameter | PKPL1P | Listing of Tenofovir (TFV) Plasma Pharmacokinetic Parameters<br>Based on Actual Time by Treatment | | SAC |
| 36. | PK<br>Parameter | PKPL1P | Listing of Emtricitabine (FTC) Plasma Pharmacokinetic Parameters Based on Actual Time by Treatment | | SAC |
| 37. | PK<br>Parameter | PKPL1P | Listing of GSK3640254 Plasma Pharmacokinetic Parameters Based on Actual Time by Treatment | | SAC |